CLINICAL TRIAL: NCT03855982
Title: Monitoring Drug-induced Myocarditis
Brief Title: Monitoring Drug-induced Myocarditis (CardiTOX)
Acronym: CardiTOX
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Assistant director, clinical investigation center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-19-03
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Myocarditis; Myocardial Failure; Myocardial Dysfunction
Keywords: myocardial toxicity; chemotherapies; drugs
MeSH Terms: conditions — Myocarditis; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- myocarditis induced by drugs and chemotherapies: Case reported in the World Health Organization (WHO) of myocarditis of patient treated by a drug, with a chronology compatible with the drug toxicity
  Interventions: Drug: Drug inducing myocarditis

INTERVENTIONS:
Drug: Drug inducing myocarditis — Drugs susceptible to induce myocarditis

SUMMARY:
Several drugs and chemotherapies seem to induce myocarditis. This study investigates reports of myocarditis, including the International classification of disease ICD-10 for treatments in the World Health Organization (WHO) global Individual Case Safety Report (ICSR) database (VigiBase).

DETAILED DESCRIPTION:
Several drugs and chemotherapies seem to have an impact on the myocardium and are responsible of myocarditis. Those are poorly described, due to the modification of the pharmacopeia, and the recent recognition of several of these adverse events. This study investigates the main characteristics of patients affected by myocarditis side effect imputed to drugs. A causality assessment according to the WHO-UMC (World Health Organization - Uppsala Monitoring Center) is systematically applied.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the WHO's pharmacovigilance database till 25/02/2019

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with a drug that could be reported in the WHO's pharmacovigilance database
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Number of myocarditis induced by drugs and report of cases of myocarditis associated with drugs. | Case reported in the World Health Organization (WHO) database of individual safety case reports to 25/02/2019

SECONDARY OUTCOMES:
Causality assessment of reported myocarditis events according to the WHO system | Case reported in the World Health Organization (WHO) database of individual safety case reports to 25/02/2019
Description of the myocarditis depending on the category of drug | Case reported in the World Health Organization (WHO) database of individual safety case reports to 25/02/2019
Description of the other related adverse events concomitant to the myocarditis induced by drugs | Case reported in the World Health Organization (WHO) database of individual safety case reports to 25/02/2019
Description of the duration of treatment when the toxicity happens (role of cumulative dose) | Case reported in the World Health Organization (WHO) database of individual safety case reports to 25/02/2019
Description of the drug-drug interactions associated with adverse events | Case reported in the World Health Organization (WHO) database of individual safety case reports to 25/02/2019
Description of the population of patients having myocarditis adverse event | Case reported in the World Health Organization (WHO) database of individual safety case reports to 25/02/2019
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed | Case reported in the World Health Organization (WHO) database of individual safety case reports to 25/02/2019

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided